CLINICAL TRIAL: NCT03120299
Title: The Effect of Omega-3 Fatty Acids on Hypertriglyceridemia in Patients With Type 2 Diabetes Mellitus
Brief Title: The Effect of Omega-3 FA on Hypertriglyceridemia in Patients With T2DM(OCEAN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCMED-20160601
Record Dates: First submitted 2017-04-15; First posted 2017-04-19 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes Mellitus; Hypertriglyceridemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertriglyceridemia | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Drug (Experimental): Omega-3 fatty acids capsules, 1 gram gel capsule, 2 capsules orally administered twice a day for 12 weeks
  Other Names:
  Omega-3 Fatty Acid fish oil Omega 3 Treasure
  Interventions: Drug: Omega-3 fatty acid
- Group B Drug (Placebo Comparator): Matching placebo capsules, 1 gram gel capsule, 2 capsules orally administered twice a day for 12 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Omega-3 fatty acid — Omega-3 fatty acids capsules, 1 gram gel capsule, 2 capsules orally administered twice a day for 12 weeks
  Other Names: fish oil supplement
  Arms: Group A Drug
Drug: Placebos — Matching placebo capsules, 1 gram gel capsule, 2 capsules orally administered twice a day for 12 weeks
  Arms: Group B Drug

SUMMARY:
The purpose of this study is to conduct a multicenter randomized, double-blind, placebo-controlled clinical trial, evaluating the effects and change of lipid metabolism, especially of triglyceride after omega-3 administration in type 2 diabetes patients with hypertriglyceride.

DETAILED DESCRIPTION:
In the present study, patients with type 2 diabetes and hypertriglyceride will be enrolled from multiple centers in China. Randomization was computer generated and stratified by center. After screening, eligible subjects will be randomly assigned into one of the following two groups: Omega-3 fatty acids capsules ( 2pills bid) and placebo capsules (2pills bid).

Blood, feces and urine samples will be collected before and after treatment. Triglycerides (TG), total cholesterol (TC), LDL-C, HDL-C, HbA1C, fasting plasma glucose (FPG), postprandial plasma glucose (PPG) will be measured. Blood metabolomics profiles of lipids, amino acids, bile acids, the change of gut microbiota, and pharmacogenomic components and parameters will be evaluated too.

Sample Size Calculation:

The primary clinical endpoint involves comparing changes in triglyceride (TG) levels between the placebo group and the omega-3 treatment group after a 12-week intervention. According to literature reports [Borthwick L J. The effects of an omega-3 ethyl ester concentrate on blood lipid concentrations in patients with hyperlipidaemia[J]. Clinical drug investigation, 1998, 15(5): 397-404], following 12 weeks of n-3 or placebo-controlled treatment, patients with hypertriglyceridemia exhibited a 9.1±24.8% increase in the placebo group and a 28.3±19.1% decrease in the omega-3 treatment group (4g/day). Based on this data, we conservatively estimate no change in TG in the placebo group for this trial, while anticipating a 10% reduction in the omega-3 treatment group. With a combined standard deviation (SD) of 30%, α=0.05, β=0.2, we calculate the sample size based on the mean difference between the two groups, resulting in N1=N2=143 cases.

Taking into account actual follow-up rates from preliminary research, we adjusted the estimated dropout rate from 20% to 5% and recalculated the sample size. Consequently, we plan to enroll 300 cases, with 150 in each of the omega-3 treatment and placebo groups, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed type 2 diabetes defined as WHO (1999) diagnostic criteria ; Both Genders Eligible;
2. Men or women aged 20 to 75 years;
3. Stable dosage of oral anti-diabetic medicine ,stable glycemia control(HbA1c<7.5%), unchanged antidiabetic therapy during the trial;
4. Hypertriglycerides (3.4mmol/L≤mean fasting blood triglycerides<22.60mmol/L, and not receiving any lipid lowering therapy for 3 days continuously or accumulated 7 days within 6 weeks before screening).

Exclusion Criteria:

1. Uncontrolled blood pressure (defined as systolic blood pressure>180mmHg or diastolic blood pressure>100mmHg);
2. Other diseases affecting lipid and glucose metabolism: hyperthyroidism，cushing syndrome ect;
3. Receiving insulin treatment in 6 months before recruitment;
4. Diagnosed heart failure, defined as New York Heart Association class III or IV;
5. Histories of acute or chronic pancreatitis，or cholelithiasis （except those received cholecystectomy）
6. Significant impaired liver function (defined as alanine transaminase (ALT)> 3 times upper limit of normal), or active liver disease;
7. PLT<60×10^9/L，Hb<100g/L；
8. Impaired renal function (defined as serum creatinine> 135 mmol/L（1.5 mg/dL, male) and > 110 mmol/L （1.3 mg/dL,female）；
9. Recorded history of malignant tumor in the past 2 years;
10. Histories of acute cerebrovascular accident within 6 months;
11. Pregnancy;
12. Known history of allergy to fish, shellfish and omega-3 fatty acids, or ineffective treatment of omega-3 fatty acids;
13. Simultaneous participation in any other clinical trial of an active pharmacologic agent within 30 days;
14. Other situations that interfere with the subject's ability to comply with study instructions;
15. Any other condition that investigators believe would interfere with the subject's ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Change in serum triglycerides from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure the serum triglycerides in blood samples before and after treatment.
Change in blood metabolomics profile of lipid species from baseline | 12 weeks
  With aid of LC/MS and GC/MS, the investigators will measure blood metabolomics profile of lipid species before and after treatment. The metabolomics measurement will help to detect the profile of all kinds of lipids species. The composition change of all these biological molecular induced by the treatment is our major interest rather than single molecular quantification.

SECONDARY OUTCOMES:
Change in serum metabolomics profile of bile acids from baseline | 12 weeks
  With aid of LC/MS and GC/MS technique, the investigators will measure the blood metabolomics molecular profile of bile acids in blood samples before and after treatment.
Change in serum metabolomics profile of amino acid species from baseline | 12 weeks
  With aid of LC/MS and GC/MS technique, the investigators will measure the blood metabolomics molecular profile of amino acid species before and after treatment.
Change in Gut microbiome from baseline | 12 weeks
  With aid of quantitative real-time PCR technique, the investigators will measure gut microbiome in fecal samples before and after treatment.
Change in fasting glucose levels from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure fasting glucose levels before and after treatment.
Change in 2-hour postprandial glucose levels from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure the 2-hour postprandial glucose levels before and after treatment.
Change in HbA1c from baseline | 12 weeks
  With aid of HPLC technique, the investigators will measure the HbA1c levels before and after treatment.
Change in Non-HDL-C from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure the non-HDL-c levels before and after treatment.
Change in serum total Cholesterol from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure serum total cholesterol levels before and after treatment.
Change in serum VLDL-c from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure serum VLDL-c levels before and after treatment.
Change in serum HDL-c from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure serum HDL-c levels before and after treatment.
Change in serum LDL-c from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure serum LDL-c levels before and after treatment.
Change in LDL-C/HDL-C from baseline | 12 weeks
  The LDL-C/HDL-C will be calculated by the ratio of the LDL-C divided by HDL-C before and after treatment.
Change in serum Apo B from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure serum Apo B levels before and after treatment.
Change in serum AST from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure serum AST levels before and after treatment.
Change in serum ALT from baseline | 12 weeks
  In aid of autoanalyser, the investigators will measure serum ALT levels before and after treatment.
Change in serum inflammation markers from baseline | 12 weeks
  With aid of autoanalyser, the investigators will measure hs-CRP, TNF-alfa, IL-6, and IL-8 etc before and after treatment.
Change in liver fat content from baseline | 12 weeks
  With aid of ultrasonic diagnostic apparatus, the investigators will measure the fat content in liver before and after treatment.
Change in Ankle-Brachial Index from baseline | 12 weeks
  The ABI value will be measured by PWV/ABI-form device (OMRON Colin Medical Instruments) before and after treatment.
Change in Brachial-ankle pulse wave velocity from baseline | 12 weeks
  The baPWV value will be measured by PWV/ABI form device (OMRON Colin Medical Instruments) before and after treatment.
Change in enrichment of fish oil in red blood cell from baseline | 12 weeks
  With aid of HPLC-ESI-MS/MS, the investigators will measure the enrichment of fish oil in red blood cell before and after treatment
Pharmacogenomics analysis | 12 weeks
  With aid of blood DNA genotyping，the investigators will compare the genotype of FASD1,FASD2 and other lipid related candidate genes with the lipid lowering effect of omega-3

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD, PHD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Lu J, Liu R, Ren H, Wang S, Hu C, Shi Z, Li M, Liu W, Wan Q, Su Q, Li Q, Zheng H, Qu S, Yang F, Ji H, Lin H, Qi H, Wu X, Wu K, Chen Y, Xu Y, Xu M, Wang T, Zheng J, Ning G, Zheng R, Bi Y, Zhong H, Wang W. Impact of omega-3 fatty acids on hypertriglyceridemia, lipidomics, and gut microbiome in patients with type 2 diabetes. Med. 2025 Jan 10;6(1):100496. doi: 10.1016/j.medj.2024.07.024. Epub 2024 Aug 19. PMID 39163858